CLINICAL TRIAL: NCT03814460
Title: Stroke and Myotonometer: Validity, Reliability and Discrimination Between the Mechanical and Sensory Component of Spasticity
Brief Title: Stroke and Assessment of Muscle Tone
Status: Completed | Type: Observational
Sponsor: University of Seville (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other); Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, Assistant Professor. Physiotherapy Department, University of Seville
Other Study IDs: Myoton18
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Muscle Tone Abnormalities; Pain; Muscle Spasticity
Keywords: Topographical mapping; Muscle state of tension; Myotonometer; Pressure Pain Threshold; Muscle Thickness
MeSH Terms: conditions — Stroke; Pain; Muscle Spasticity | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: A control group of healthy subjects with no previous history of neurological disorders or conditions. This group pf participants will be selected in a similar population based-cohort than the other two study groups.
  Interventions: Diagnostic Test: Assessment of Tone, Pain and Thickness
- Acute Stroke Group: In this group, participants who suffered a previous stroke within 3 months before data collection will be included.
  Interventions: Diagnostic Test: Assessment of Tone, Pain and Thickness
- Chronic Stroke Group: In this group, only participants who have suffered a previous stroke of more than 3 months duration before data collection will be included.
  Interventions: Diagnostic Test: Assessment of Tone, Pain and Thickness

INTERVENTIONS:
Diagnostic Test: Assessment of Tone, Pain and Thickness — Evaluation of Muscle state of tension, self-reported response to mechanical pressure pain and muscle thickness. The evaluation process of muscle tone and pressure pain sensitivity will be carried out following a topographical mapping covering myotendinous and muscle belly sites in the biceps brachii and the gastrocnemius muscles

SUMMARY:
Spasticity is defined as a state of increased muscle tone, which evokes an increased resistance to a passive and fast stretching of the muscle. Indeed, the degree of spasticity depends, among other things, on the stretching velocity performed to the muscle. However, most of the tools used in the clinical setting to assess spasticity do not take into account the relationship between increased muscle tone and speed of stretching. Instead of that, muscle tone is usually assessed in a relaxed position of the muscle.

Likewise, to date, despite the functional disabilities related to the presence of chronic pain after a stroke, no previous study has correlated muscle tone and pressure pain sensitivity within this population

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years
* Clinical diagnosis of stroke, confirmed using a MRI.
* No previous history of other strokes.
* Increases muscle tone in upper and lower extremities (punctuation equal to or superior to 1 in the Tardieu Scale, Ashworth Scale)
* Ability to understand the study goals, follow simple instructions and provide informed consent.
* Score equal to or superior to 24 in the Minimental State Examination.

Exclusion Criteria:

* Any other confirmed neurological disorder that may influence muscle tone (multiple sclerosis, Parkinson, muscle dystrophies...)
* A chronic musculoskeletal disorder in the upper or lower limb.
* Previous history of surgery in the upper or lower extremities.
* Changes in the medication intake that may affect muscle tone assessments in the 48 hours before data collection.
* Having received botulin toxin in gastrocnemius or biceps brachii muscles in the 30 days before data collection.
* A concomitant acute infection during data collection.
* A previous epileptic crisis in the week before the study or during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with acute or chronic stroke will be recruited from large public hospitals. The control participants will be selected from the same population-based cohort
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold, assessed by Manual Pressure Algometry | One time assessment
  A handheld electronic pressure algometer with a 1-cm2 contact probe will be used. Pressure pain thresholds (PPTs), as the minimum necessary pressure force to evoke pain, will be assessed bilaterally over biceps brachii and the gastrocnemius muscles (medial and lateral). Assessments will be made using a topographical mapping covering myotendinous and muscle belly sites in the above mentioned muscles. A 30-second break will be used between assessments to prevent bruising, and an average of the two measures over each site will be calculated for the statistical analysis. Pressure algometry is reliable in healthy individuals, and in stroke patients
Muscle Tone Assessment, using the modified Tardieu Scale | One time assessment
  The modified Tardieu Scale is the most common tool used in the clinical setting to evaluate the muscle tone. The muscle response to a slow and fast stretching will be performed. During the fast stretching, the joint angle in which the muscle responds with difficulty will be collected using an electrogoniometer.

SECONDARY OUTCOMES:
Muscle Stiffness, assessed by a myotonometer | One time assessment
  The stiffness of the biceps brachii and gastrocnemius muscles will be collected using a handheld myotonometer device, the so-called MyotonPRO, (Myoton AS, Estonia). The MyotonPRO is small, non-invasive, and it has shown good validity and high reliability in larger and smaller body muscles. This device delivers a multi-scan mode of three brief mechanical impulses, each one shortly followed by a quick release, to record the damped natural oscillation of the muscle using an accelerometer.
  Evaluations will be made in the affected and non-affected sides of stroke patients and in dominant and non-dominant sides of control participants.
Muscle State of Tension (Muscle Tone), assessed by a myotonometer | One time assessment
  The tone of the biceps brachii and gastrocnemius muscles will be collected using a handheld myotonometer device, the MyotonPRO, (Myoton AS, Estonia). The MyotonPRO is small, non-invasive, and it has shown good validity and high reliability in larger and smaller body muscles. This device delivers a multi-scan mode of three brief mechanical impulses, each one shortly followed by a quick release, to record the damped natural oscillation of the muscle using an accelerometer.
  Evaluations will be made in the affected and non-affected sides of stroke patients and in dominant and non-dominant sides of control participants.
Muscle Thickness | One time assessment
  The thickness of the assessed muscles will be evaluated using ecography. Muscle thickness will be assessed in one point corresponding to a myotendinous site and one point corresponding to a muscle belly location in both, the biceps brachii and gastrocnemius muscles.
  Evaluations will be made in the affected and non-affected sides of stroke patients and in dominant and non-dominant sides of control participants.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Garcia Bernal, PT, Principal Investigator — Physiotherapy Department, University of Sevilla, Spain
Locations (2):
- Spain (2):
  - Physiotherapy Department, University of Seville, Seville
  - University of Sevilla, Seville

IPD SHARING:
Plan to Share IPD: Undecided